CLINICAL TRIAL: NCT00700063
Title: A Multicenter, Randomized, Double-blind, Vehicle-controlled, Dose-ranging Study to Evaluate the Safety and Efficacy of 0.005%, 0.01% and 0.015% PEP005 Topical Gel When Used to Treat Actinic Keratoses on the Head (Face or Scalp)
Brief Title: A Multicenter Study to Evaluate the Safety and Efficacy of PEP005 Topical Gel When Used to Treat Actinic Keratoses on the Head (Face or Scalp)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peplin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEP005-015
Record Dates: First submitted 2008-06-15; First posted 2008-06-18 (Estimated); Results first posted 2012-08-22 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Actinic Keratosis
Keywords: Peplin; Actinic keratosis; PEP005
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 1 (Experimental)
  Interventions: Drug: PEP005 Topical Gel
- 2 (Experimental)
  Interventions: Drug: PEP005 Topical Gel
- 3 (Experimental)
  Interventions: Drug: PEP005 Topical Gel
- 4 (Placebo Comparator)
  Interventions: Drug: Vehicle gel
- 5 (Experimental)
  Interventions: Drug: PEP005 Topical Gel
- 6 (Experimental)
  Interventions: Drug: PEP005 Topical Gel
- 7 (Experimental)
  Interventions: Drug: PEP005 Topical Gel
- 8 (Placebo Comparator)
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: PEP005 Topical Gel — 0.005%, two days treatment
  Arms: 1
Drug: PEP005 Topical Gel — 0.01%, two days treatment
  Arms: 2
Drug: PEP005 Topical Gel — 0.015%, two days treatment
  Arms: 3
Drug: Vehicle gel — two days treatment
  Arms: 4
Drug: PEP005 Topical Gel — 0.005%, three days treatment
  Arms: 5
Drug: PEP005 Topical Gel — 0.01%, three days treatment
  Arms: 6
Drug: PEP005 Topical Gel — 0.015%, three days treatment
  Arms: 7
Drug: Vehicle gel — three days treatment
  Arms: 8

SUMMARY:
This Phase IIb study is designed to assess the safety and efficacy of 0.005%, 0.01% and 0.015% PEP005 Topical Gel when applied to an area of skin, containing 4-8 AK lesions on the face or scalp.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or female
* Female patients must be of
* Non-childbearing potential;
* Childbearing potential, provided negative pregnancy test and using effective contraception
* 4 to 8 AK lesions on the face or scalp

Exclusion Criteria:

* Cosmetic or therapeutic procedures within 2 weeks and within 2 cm of the selected treatment area.
* Treatment with immunomodulators, or interferon/ interferon inducers or systemic medications that suppress the immune system: within 4 weeks.
* Treatment with 5-FU, imiquimod, diclofenac, or photodynamic therapy:

within 8 weeks and 2 cm of treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (25):
  - Burke Pharmaceutical Research, Hot Springs, Arizona
  - Dermatology Research of Arkansas, Little Rock, Arkansas
  - Koppel Dermatology, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Integrated Research Group Inc, Riverside, California
  - Skin Surgery Medical Group Inc, San Diego, California
  - 470 Castro St Suite 202-204, San Francisco, California
  - Solano Clinical Research, Vallejo, California
  - Dermatology Specialists Inc, Vista, California
  - Spencer Derm and Skin Surgery Center, St. Petersburg, Florida
  - Northwest Clinical Trial, Boise, Idaho
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Christie Clinic, Champaign, Illinois
  - South Bend Clinic, South Bend, Indiana
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - TKL Research, Inc., Paramus, New Jersey
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Oregon Medical Research Center, Portland, Oregon
  - Philadelphia Institute of Dermatology, Philadelphia, Pennsylvania
  - Dermatology Research Associates, Nashville, Tennessee
  - DermResearch, Inc. 8140 N. MoPac, Bldg. 3, Suite 120,, Austin, Texas
  - Suzanne Bruce and Associates, The Center for Skin Research, Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Dermatology Associates of Tyler, Tyler, Texas
- Australia (3):
  - Southderm Pty Ltd, Kogarah, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Siller Medical, Brisbane, Queensland

REFERENCES:
- See also: Food and Drug Authority — http://www.fda.gov/
- See also: Therapeutic Goods Administration — http://www.tga.gov.au/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient randomized: 24 June 2008 Last patient completed Day 57: 20 October 2008
Groups:
- 1. PEP005 Topical Gel 0.005%; 3. PEP005 Topical Gel 0.015%: Two days treatment day 1, 2
- 2. PEP005 Topical Gel 0.01%; 4. Vehicle Gel: Two days treatment, day 1, 2
- 5. PEP005 Topical Gel 0.005%; 6. PEP005 Topical Gel 0.01%; 7. PEP005 Topical Gel 0.015%; 8. Vehicle Gel: Three days treatment, day 1, 2, 3
Period: Overall Study
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Started | 33 | 34 | 33 | 33 | 33 | 34 | 32 | 33
Completed | 32 | 34 | 33 | 31 | 31 | 34 | 32 | 33
Not Completed | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel | Total
Number analyzed (Participants) | 33 | 34 | 33 | 33 | 33 | 34 | 32 | 33 | 265
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 13 | 16 | 18 | 11 | 13 | 14 | 11 | 112
  >=65 years | 17 | 21 | 17 | 15 | 22 | 21 | 18 | 22 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (10.2) | 67.5 (10.5) | 67.8 (7.0) | 65.2 (9.7) | 68.7 (11.0) | 67.7 (9.0) | 67.2 (10.1) | 69.3 (10.7) | 67.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 4 | 6 | 3 | 4 | 5 | 28
  Male | 30 | 32 | 32 | 29 | 27 | 31 | 28 | 28 | 237
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 31 | 29 | 29 | 31 | 25 | 28 | 232
  Australia | 3 | 5 | 2 | 4 | 4 | 3 | 7 | 5 | 33

OUTCOME MEASURES:

1. Primary Outcome: Incidence of AEs Recorded Throughout the Study
Description: Incidence of AEs recorded throughout the study
Time Frame: 57 days
Population: One patient in the PEP005 Topical Gel 0.005% group received no dose of study medication and were therefore not included in the safety population.
Measure: Number; unit: participants
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Number analyzed (Participants) | 32 | 34 | 33 | 33 | 33 | 34 | 32 | 33
participants | 12 | 12 | 8 | 11 | 11 | 14 | 22 | 6

2. Secondary Outcome: Efficacy (Clearance of AK Lesions) Partial Clearance Rate
Description: Partial clearence rate, defined as the number of patients at the Day 57 visit with a 75% or greater reduction in the number of AK lesions identified at baseline, in the Face and Scalp
Time Frame: 57 days
Measure: Number; unit: participants
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Number analyzed (Participants) | 33 | 34 | 33 | 33 | 33 | 34 | 32 | 33
participants | 11 | 17 | 17 | 3 | 14 | 9 | 23 | 4

3. Primary Outcome: Incidence of SAE Recorded Throughout the Study
Description: Incidence of SAE recorded throughout the study
Time Frame: 57 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Number analyzed (Participants) | 32 | 34 | 33 | 33 | 33 | 34 | 32 | 33
participants | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

4. Primary Outcome: Incidence Rate and Severity of LSRs Following Study Medication Application
Description: The treatment area was assessed at baseline, Day 1 (pre-dose), and at each subsequent study visit for the presence and grade (0 to 4) of the following LSRs: erythema; flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration. A composite LSR score (0 to 24), reflecting the sum of each individual LSR grade, was calculated for each patient at each visit.
  The actual value and change from baseline in the composite LSR score were also summarized.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Number analyzed (Participants) | 32 | 34 | 33 | 33 | 33 | 34 | 32 | 33
scores on a scale | 1.4 (1.3) | 1.6 (1.3) | 1.3 (0.9) | 1.4 (1.1) | 1.6 (1.5) | 1.5 (1.3) | 1.3 (1.0) | 1.7 (1.2)

5. Primary Outcome: Incidence Rate and Severity of LSRs Following Study Medication Application
Description: as for outcome 4
Time Frame: Day 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Number analyzed (Participants) | 32 | 34 | 33 | 33 | 33 | 34 | 32 | 33
units on a scale | 0.8 (1.1) | 1.1 (1.0) | 0.8 (0.8) | 1.3 (1.2) | 1.4 (1.4) | 1.1 (1.0) | 0.8 (1.3) | 1.1 (0.9)

6. Primary Outcome: Incidence of Hyperpigmentation Following Study Medication Application
Description: The selected treatment area was assessed for hyperpigmentation at baseline (Day 1 pre-dose), Day 57, and at each poststudy followup visit as warranted.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Number analyzed (Participants) | 32 | 34 | 33 | 33 | 33 | 34 | 32 | 33
participants | 15 | 15 | 11 | 8 | 13 | 12 | 15 | 15

7. Primary Outcome: Incidence of Hyperpigmentation Following Study Medication Application
Description: The selected treatment area was assessed for hyperpigmentation at baseline (Day 1 pre-dose), Day 57, and at each poststudy followup visit as warranted. If any pigmentation was present, the significance and extent of pigmentation and scarring was recorded. At all timepoints, pigmentation evaluations were performed by a board certified Dermatologist (or equivalent)
Time Frame: Day 57
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Number analyzed (Participants) | 32 | 34 | 33 | 33 | 33 | 34 | 32 | 33
participants | 13 | 13 | 7 | 6 | 8 | 11 | 11 | 15

8. Primary Outcome: Incidence of Hypopigmentation Following Study Medication Application
Description: The selected treatment area was assessed for hypopigmentation at baseline (Day 1 pre-dose), Day 57, and at each poststudy followup visit as warranted. If any pigmentation was present, the significance and extent of pigmentation and scarring was recorded. At all timepoints, pigmentation evaluations were performed by a board certified Dermatologist (or equivalent)
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Number analyzed (Participants) | 32 | 34 | 33 | 33 | 33 | 34 | 32 | 33
participants | 7 | 10 | 6 | 8 | 10 | 9 | 16 | 6

9. Primary Outcome: Incidence of Hypopigmentation Following Study Medication Application
Description: as for outcome 8
Time Frame: Day 57
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Number analyzed (Participants) | 32 | 34 | 33 | 33 | 33 | 34 | 32 | 33
participants | 4 | 6 | 6 | 6 | 9 | 9 | 12 | 6

10. Primary Outcome: Incidence of Scarring Following Study Medication Application
Description: The selected treatment area was assessed for scarring at baseline (Day 1 pre-dose), Day 57, and at each poststudy followup visit as warranted. If any scarring was present, the significance and extent of scarring was recorded. At all timepoints, pigmentation evaluations were performed by a board certified Dermatologist (or equivalent)
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Number analyzed (Participants) | 32 | 34 | 33 | 33 | 33 | 34 | 32 | 33
participants | 1 | 3 | 2 | 3 | 6 | 1 | 10 | 3

11. Primary Outcome: Incidence of Scarring Following Study Medication Application
Description: as for outcome 10
Time Frame: Day 57
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Number analyzed (Participants) | 32 | 34 | 33 | 33 | 33 | 34 | 32 | 33
participants | 1 | 1 | 1 | 1 | 5 | 1 | 5 | 2

12. Primary Outcome: Complete Clearance Rate of AK Lesions;
Description: Defined as the number of patients at the day 57 post-treatment visit with no clinically visible AK lesions in the selected treatment area
Time Frame: Day 57
Measure: Number; unit: participants
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Number analyzed (Participants) | 33 | 34 | 33 | 33 | 33 | 34 | 32 | 33
participants | 5 | 10 | 12 | 0 | 11 | 6 | 16 | 3

ADVERSE EVENTS:
Time Frame: 57 days
Description: One patient in the PEP005 Topical Gel 0.005% group received no dose of study medication and were therefore not included in the safety population.
Arm/Group | 1. PEP005 Topical Gel 0.005% | 2. PEP005 Topical Gel 0.01% | 3. PEP005 Topical Gel 0.015% | 4. Vehicle Gel | 5. PEP005 Topical Gel 0.005% | 6. PEP005 Topical Gel 0.01% | 7. PEP005 Topical Gel 0.015% | 8. Vehicle Gel
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/34 | 0/33 | 0/33 | 1/33 | 0/34 | 1/32 | 0/33
Other Adverse Events (participants affected / at risk) | 8/32 | 5/34 | 5/33 | 3/33 | 7/33 | 8/34 | 12/32 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. PEP005 Topical Gel 0.005% (N=32) | 2. PEP005 Topical Gel 0.01% (N=34) | 3. PEP005 Topical Gel 0.015% (N=33) | 4. Vehicle Gel (N=33) | 5. PEP005 Topical Gel 0.005% (N=33) | 6. PEP005 Topical Gel 0.01% (N=34) | 7. PEP005 Topical Gel 0.015% (N=32) | 8. Vehicle Gel (N=33)
gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1. PEP005 Topical Gel 0.005% (N=32) | 2. PEP005 Topical Gel 0.01% (N=34) | 3. PEP005 Topical Gel 0.015% (N=33) | 4. Vehicle Gel (N=33) | 5. PEP005 Topical Gel 0.005% (N=33) | 6. PEP005 Topical Gel 0.01% (N=34) | 7. PEP005 Topical Gel 0.015% (N=32) | 8. Vehicle Gel (N=33)
APPLICATION SITE IRRITATION (General disorders) | 3 | 3 | 4 | 1 | 2 | 3 | 7 | 0
APPLICATION SITE PRURITUS (General disorders) | 3 | 3 | 0 | 0 | 4 | 5 | 1 | 0
APPLICATION SITE DISCOMFORT (General disorders) | 1 | 1 | 0 | 0 | 3 | 0 | 2 | 0
APPLICATION SITE SWELLING (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
APPLICATION SITE PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
APPLICATION SITE INFECTION (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
NASOPHARYNGITIS (Infections and infestations) | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0
EYELID OEDEMA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and Investigator agree not to publish the results of this study without the prior written consent of Sponsor. As used herein, the term 'publish' shall include oral presentations, written abstracts, written manuscripts, etc.